CLINICAL TRIAL: NCT05286229
Title: A Phase 1 Study to Evaluate the Safety, Tolerability and Pharmacokinetics of Etentamig (ABBV-383) Monotherapy in Japanese Subjects With Relapsed or Refractory Multiple Myeloma (4L+ RRMM Monotherapy Study)
Brief Title: A Study to Assess Adverse Events and Change in Disease State of Intravenously (IV) Infused Etentamig (ABBV-383) of Adult Participants With Relapsed or Refractory Multiple Myeloma in Japan
Status: Active, not recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: AbbVie (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: M22-984
Record Dates: First submitted 2022-03-17; First posted 2022-03-18 (Actual); Last update posted 2025-08-08 (Actual); Status verified 2025-08

CONDITIONS: Relapsed/Refractory Multiple Myeloma
Keywords: Relapsed/Refractory Multiple Myeloma; Etentamig; Cancer
MeSH Terms: conditions — Multiple Myeloma; Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Cohort 1 (Etentamig Dose A) (Experimental): Participants with relapsed or refractory (R/R) multiple myeloma (MM) who meet the criteria outline in the protocol will receive Etentamig Dose A in 21-day cycles.
  Interventions: Drug: Etentamig
- Cohort 2 (Etentamig Dose B) (Experimental): Participants with R/R MM who meet the criteria outline in the protocol will receive Etentamig Dose B in 21-day cycles.
  Interventions: Drug: Etentamig

INTERVENTIONS:
Drug: Etentamig — Intravenous (IV) Infusion

SUMMARY:
Multiple myeloma (MM) is an incurable disease characterized by the growth of monoclonal plasma cells in the bone marrow. The purpose of this study is to assess the adverse events and change in disease state of etentamig in adult participants with relapsed/refractory (R/R) multiple myeloma (MM). Adverse events and change in disease state will be assessed.

Etentamig (ABBV-383) is an investigational drug being developed for the treatment of R/R MM. Study doctors put the participants in groups called treatment arms. Two doses of ABBV-383 will be explored. Each treatment arm receives a different dose of ABBV-383 to determine a tolerable dose. Approximately 12 adult participants with R/R MM will be enrolled in the study in approximately 6 sites in Japan.

Participants will receive intravenous (IV) Etentamig (ABBV-383) at two increasing doses in 21-day cycles.

There may be higher treatment burden for participants in this trial compared to their standard of care. Participants will attend regular visits during the study at an approved institution (hospital or clinic). The effect of the treatment will be frequently checked by medical assessments, blood tests, and and monitoring of side effects.

ELIGIBILITY:
Inclusion Criteria:

* Eastern Cooperative Oncology Group (ECOG) performance of <= 2.
* Must have adequate bone marrow function as defined in the protocol.
* Must meet laboratory parameters as outlined in the protocol.
* Must have a confirmed diagnosis of relapsed/refractory (R/R) multiple myeloma (MM) with documented evidence of progression during or after the participant's last treatment regimen based on the investigator's determination of the International Myeloma Working group (IMWG) criteria.

  * Relapsed defined as previously treated myeloma that progresses and requires initiation of salvage therapy, but does not meet criteria for refractory myeloma.
  * Refractory defined as disease that is nonresponsive (failure to achieve minimal response or development of progressive disease) while on primary or salvage therapy, or progresses within 60 days of last therapy.
* Must have received at least 3 prior lines of therapy (including exposure to a proteasome inhibitor (PI), an immunomodulatory imide (IMiD), and an anti-CD38 mAb).
* Must have measurable disease within 28 days of enrollment, defined as at least 1 of the following:

  * Serum M-protein >= 0.5 g/dL (>= 5 g/L).
  * Urine M-protein >= 200 mg/24 hours.
  * Serum free light chain (FLC) >= 100 mg/L (involved light chain) and an abnormal serum kappa lambda ratio only for participants without measurable serum or urine M-protein.
* Consents to a fresh pretreatment bone marrow tumor biopsy or has adequate archival bone marrow tumor tissue that was collected within 12 weeks prior to screening and without intervening treatment.

Exclusion Criteria:

- Has received B-cell maturation antigen (BCMA)-targeted therapy. Participants who have received targeted therapy against non-BCMA targets will not be excluded.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 8 (Actual)
Dates: Start 2022-03-24 (Actual); Primary Completion 2026-03 (Estimated); Study Completion 2026-03 (Estimated)

PRIMARY OUTCOMES:
Number of Dose-Limiting Toxicities (DLT) | Up to Approximately 12 Months
  DLT events are defined as adverse events or abnormal laboratory values assessed as "reasonable possibility" of relationship to the administration of Etentamig, which cannot be attributed by the investigator to a clearly identifiable cause such as disease progression or concurrent illness.
Number of Participants with Adverse Events (AE) | Up to Approximately 24 Months
  AE is defined as any untoward medical occurrence in a participant or clinical investigation participant administered a pharmaceutical product and which does not necessarily have a causal relationship with this treatment.

SECONDARY OUTCOMES:
Objective Response Rate (ORR) | Up to Approximately 24 Months
  ORR is defined as the percentage of participants who achieve confirmed partial response (PR) or better determined by International Myeloma Working Group (IMWG) criteria, prior to the initiation of subsequent myeloma therapy.
Progression Free Survival (PFS) | Up to Approximately 24 Months
  PFS is defined as the duration from the date of first dose to the date of disease progression (PD) determined by IMWG criteria, or death, whichever occurs first.
Time to Response (TTR) | Up to Approximately 24 Months
  TTR is defined as the number of months from the date of first dose to the date of best overall response of CR or PR ('responders') determined by IMWG criteria as assessed by investigator.
Duration of Response (DOR) | Up to Approximately 24 Months
  DOR is defined as the number of days from the day the response criteria are met to the date that disease progression is objectively documented.
Minimal Residual Disease (MRD) Negativity Rate | Up to Approximately 24 Months
  MRD is defined as the percentage of participants with assessment of the minimal residual disease negativity.

CONTACTS AND LOCATIONS:
Overall Officials: ABBVIE INC., Study Director — AbbVie
Locations (6):
- Japan (6):
  - National Cancer Center Hospital East /ID# 240943, Kashiwa-shi, Chiba
  - Hokkaido University Hospital /ID# 242672, Sapporo, Hokkaido
  - Kanazawa University Hospital /ID# 240948, Kanazawa, Ishikawa-ken
  - Duplicate_Okayama Medical Center /ID# 240949, Okayama, Okayama-ken
  - The University of Osaka Hospital /ID# 242032, Suita-shi, Osaka
  - Yamagata University Hospital /ID# 240945, Yamagata, Yamagata

IPD SHARING:
Plan to Share IPD: No